CLINICAL TRIAL: NCT02665442
Title: Esophageal Stylet as a Strategy to Minimize the Risk of Esophageal Injury During the Atrial Fibrillation Catheter Ablation Procedure.
Brief Title: Retracting the Esophagus During AF Ablation
Acronym: EsoSure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northeast Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1511016760
Record Dates: First submitted 2016-01-23; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation; Esophageal Fistula; Cardiac Arrhythmia
Keywords: Esophageal Stylet; EsoSure; Atrial Fibrillation; Catheter Ablation; Mechanical esophageal displacement
MeSH Terms: conditions — Atrial Fibrillation; Esophageal Fistula; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stylet (Experimental): This group will receive an Esophageal stylet; EsoSure during the ablation procedure in attempt of moving the esophagus away from the ablation site.
  Interventions: Device: Esophageal Stylet - EsoSure
- Non-Stylet (No Intervention): This group will receive the ablation procedure without any modifications or interventions. No esophageal stylet will be used in this group.

INTERVENTIONS:
Device: Esophageal Stylet - EsoSure — The Esophageal Stylet is a thin rigid tube, which will be inserted inside a commonly used nasogastric tube placed inside the esophagus during the ablation. We will use this stylet to move the esophagus away from the site of the ablation about 1-2 centimeters.
  Other Names: Esophageal Retractor
  Arms: Stylet

SUMMARY:
This Study is designed to determine the outcome and effect of implementation of Esophageal Stylet as a strategy to minimize the risk of esophageal injury during the atrial fibrillation catheter ablation procedure.

DETAILED DESCRIPTION:
There is a clear potential to produce transmural esophageal injury during catheter ablation for AF when employing a lesion set targeting the posterior left atrial wall and pulmonary vein (PV) antra using contemporary large-tip or irrigated-tip catheter ablation systems when endocardial target sites are in close proximity to the esophagus.

It is very likely that a movement by the Esophageal Stylet of only 2 to 3 centimeters from the midline can safely protect the esophagus from thermal injury and will mimic the natural migration of the esophagus itself.

The Stylet proposes to safely facilitate lateral esophageal movement in a manner consistent with the esophagus's own natural migration in order to displace and maintain the esophagus's position away from potential damage resulting from a cardiac ablation procedure in the left atrium or coronary sinus.

The Esophageal Stylet is a thin rigid tube, which will be inserted inside a commonly used nasogastric tube placed inside the esophagus during the ablation. We will use this stylet to move the esophagus away from the site of the ablation about 1-2 centimeters. Other common procedures, such as (Trans-esophageal Echocardiogram), move the esophagus twice this distance with a low risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above for the Patient or legal representative to provide informed consent.
2. Documented paroxysmal or persistent Atrial Fibrillation by a Cardiologist and EKG finding.
3. The patient will undergo Atrial Fibrillation catheter ablation as a treatment plan.

Exclusion Criteria:

1. Bleeding disorder.
2. Dysphagia to solid and liquid or any documented esophageal masses or cancer.
3. Esophageal varices, diverticulum, esophageal web, upper GI bleeding, or hiatal hernia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal injury or erosion | 2-3 days post ablation
  Decrease of esophageal thermal injury detected by esophageal Pill-Cam

SECONDARY OUTCOMES:
Recurrence of Atrial Fibrillation | 12 Months
  Decrease of atrial fibrillation recurrence after 12 months
Total radiofrequency time | Day of ablation procedure
  Decrease the total time of radiofrequency ablation at the procedure time

CONTACTS AND LOCATIONS:
Overall Officials: Mark Marieb, MD, FACC, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through publications.